CLINICAL TRIAL: NCT03221114
Title: Positive Psychology Intervention for Spanish-speaking Hispanic/Latino Adults at Risk for Cardiovascular Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1K01HL130712-01A1 (NIH)
Record Dates: First submitted 2017-06-14; First posted 2017-07-18 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Uncontrolled Hypertension; Cardiovascular Risk Factor
Keywords: Hispanics/Latinos; Underserved Population

STUDY DESIGN:
Intervention Model Description: Cluster-randomized control trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blind to intervention assignment and will only collect clinical data at baseline, 8-, and 12-weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Psychological Intervention (Experimental): Our culturally-tailored Positive Psychology (PP) Intervention is a non-pharmacotherapy approach aimed at increasing positive emotional experiences by teaching individuals to engage in intentional activities known to increase psychological and emotional well-being through targeting of constructs such as optimism, gratitude, mindfulness/relaxation, and resilience.
  Interventions: Behavioral: Positive Psychological Intervention
- Wait list control (No Intervention): Receipt after the active treatment group has completed the positive psychological intervention.

INTERVENTIONS:
Behavioral: Positive Psychological Intervention — Our culturally-tailored Positive Psychology Intervention is a non-pharmacotherapy approach aimed at increasing positive emotional experiences by teaching individuals to engage in intentional activities known to increase psychological and emotional well-being through targeting of constructs such as optimism, gratitude, mindfulness/relaxation, and resilience.
  Other Names: Positive Affect Intervention
  Arms: Positive Psychological Intervention

SUMMARY:
The largest epidemiologic study of Hispanic/Latino participants thus far, i.e., the Hispanic Community Health Study/Study of Latinos (HCHS/SOL) documented that 80% of men and 71% of women have at least one major cardiovascular disease (CVD) risk factor. The American Heart Association emphasizes that current CVD prevention efforts are sparse and ineffectual in minority populations and acknowledges the need for new and more effective disease prevention strategies. This observational study and pilot cluster-randomized clinical trial seeks to implement and evaluate a novel 8-week Positive Psychology (PP) Intervention (compared to an attention control condition) in Hispanic/Latino adults with uncontrolled hypertension, i.e., elevated 24-hour ambulatory blood pressure, with primary interest in testing efficacy for clinically meaningful improvements in cardiovascular function.

DETAILED DESCRIPTION:
The study features piloting of a cluster-randomized trial to determine whether a positive psychology (PP) intervention is associated with greater improvements in blood pressure compared to an attention control condition. The pilot trial additionally evaluates the efficacy of the PP intervention with respect to psychological well-being, hypertension-related health behaviors, autonomic cardiac control, and high-sensitivity C-reactive protein. Serum blood assays will facilitate exploration of mechanistic indicators linking psychological well-being to cardiac functioning.

ELIGIBILITY:
Inclusion Criteria:

* Hispanics/Latinos recruited from Catholic church sites in Chicago-land area
* aged ≥18
* fluent in English or Spanish with ≥8th grade education
* elevated 24-hour ambulatory blood pressure levels (systolic BP> 140 mmHg and >90 mmHg for diastolic BP).

Exclusion Criteria:

* Unavailable for study period; have cognitive impairment denoting dementia
* have severely reduced life expectancy
* are currently enrolled in psychotherapy or take prescribed antidepressants
* history or current diagnosis of bipolar disorder, dissociative disorder, psychosis, or substance abuse
* have severe depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Ambulatory Blood Pressure at 8- and 12-weeks | Baseline, 8-, and 12-weeks
  The device, Vitavue, consists of a wireless microcontroller that connects to a desktop computer running proprietary software when operated in real time connected mode. Alternatively, it can be operated in standalone unconnected mode by logging acquired data to an internal memory storage device. The device contains a number of sensors including ECG single channel amplifier, Multispectral Photodiode to record photo pulse plethysmograms, temperature sensor to measure skin temperature, and an accelerometer to record the level of activity.

SECONDARY OUTCOMES:
Center for Epidemiological Studies Depression Scale (CESD): Change from Baseline Depressive Symptoms at 8- and 12-weeks | Baseline, 8-, and 12-weeks
  Center for Epidemiological Studies Depression-Scale
Life Orientation Test-Revised (LOT-R): Change from Baseline Dispositional Optimism at 8- and 12-weeks | Baseline, 8-, and 12-weeks
  Life Orientation Test-Revised
General Well-being Schedule: Change in Baseline Emotional Vitality at 8- and 12-weeks | Baseline, 8-, and 12-weeks
  General Well-being Schedule
Life Engagement Test (LET): Change in Baseline Life engagement and Meaning at 8- and 12-weeks | Baseline, 8-, and 12-weeks
  Life Engagement Test

OTHER OUTCOMES:
Physical Activity: Change in Hypertension-related Health Behavior(s) | Baseline, 8-, and 12-weeks
  Physical Activity using Fitbit One
Diet: Change in Hypertension-related Health Behavior(s) | Baseline, 8-, and 12-weeks
  Diet using Scored Sodium Questionnaire
Change in Heart Rate Variability | Baseline, 8-, and 12-weeks
  Beat-to-beat interval
Change in High-sensitivity C-Reactive Protein | Baseline, 8-, and 12-weeks
  mg/L

CONTACTS AND LOCATIONS:
Locations (1):
- St. Pius V Parish, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make the data available to users only under a data-sharing agreement that provides for: (1) a commitment to use data only for research purposes and not to identify any individual participant; (2) a commitment to secure the data using appropriate technology; and (3) a commitment to destroy or return data after analyses are completed. If additional outputs result from this research that would be appropriate to share with a wider audience, we will work with the Research Data Service at the University Library to determine appropriate venues for archiving and sharing.